CLINICAL TRIAL: NCT05980858
Title: Effects of Exogenous Ketosis on Renal Function, Renal Perfusion, and Sodium Excretory Capacity in Healthy Subjects
Acronym: KETO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TZL-2-2023
Record Dates: First submitted 2023-07-05; First posted 2023-08-08 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Ketosis; Ketonemia
Keywords: Kidney circulation; Kidney physiology; Kidney function; Glomerular Filtration Rate
MeSH Terms: conditions — Ketosis | interventions — 3-Hydroxybutyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KetoneAid KE4, then Placebo drink (Active Comparator): For five days each subject will receive beta-hydroxybutyrate (KE4), then crossed over to receive placebo drink for 5 days.
  Interventions: Dietary Supplement: Beta-hydroxybutyrate; Other: Placebo
- Placebo drink, then KetoneAid KE4 (Active Comparator): For five days each subject will receive a placebo drink three times daily, then subjects are crossed over to receive beta-hydroxybutyrate (KE4).
  Interventions: Dietary Supplement: Beta-hydroxybutyrate; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-hydroxybutyrate — Each subject receive Beta-hydroxybutyrate 300mg/kg x 3 for five days. After the treatment period effect variables will be examined.
Other: Placebo — Each subject receive a placebo drink 3 x day for five days. After the treatment period effect variables will be examined.

SUMMARY:
This is a randomized, placebo-controlled, double-blinded crossover design. Fifteen healthy subjects will be randomized to receive either ketone bodies (KE4) or placebo delivered by KetoneAid. After a period of 5-days treatment, effect variables will be measured (experiment day 1). After a washout period of 14 days, the subjects are crossed over to a similar treatment period with the other treatment. The study is terminated by measuring effect variables after the second treatment period (experiment day 2).

DETAILED DESCRIPTION:
Background: Renewed interest in ketone bodies has emerged, partly driven by the recent success of selective sodium glucose co transporter 2 (SGLT-2) inhibition in preventing cardiovascular deaths in patients with diabetes mellitus (DM) and chronic kidney disease (CKD). Effects of ketosis are of importance in order to understand the beneficial effects of SGLT-2 inhibitors and to account for the full therapeutic potential of this treatment.

Hypothesis: Ketosis increases renal blood flow and glomerular filtration rate (GFR).

Methods: It is a randomized, placebo-controlled double-blinded cross over study. Fifteen healthy subjects will be randomized to receive either ketone bodies (KE4) or for 5 days. After a wash out period of at least 14 days, the subjects are crossed over to receive the other treatment. After each treatment period effect variables will be measured including Technetium(Tc)99m - Diethylenetriamine pentaacetate (DTPA) clearance and water based positron emission tomography computed tomography (PET/CT)

Perspectives: The study has the potential to provide information regarding the therapeutic potential of treatment with ketone bodies and understanding of conditions characterized by ketosis, such as SGLT2-inhibitor treatment.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/m2
* Safe contraception if women in childbearing age
* Normal biochemical screening

Exclusion Criteria:

* Pregnancy or breast feeding
* Major heart-, liver-, kidney-, lung-, neurological- or endocrine disease
* Daily use of prescription drugs (expect for contraceptives)
* Alcohol or drug abuse
* Periodic fasting
* Routinely intake of ketogenic diet

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
GFR | Measured after each treatment period (day 6 and approximately day 26)
  Change in GFR measured by Tc99m-DTPA clearance
Renal Blood Flow (RBF) | Subjects are scanned after each treatment period (day 6 and approximately day 26)
  Change in RBF determined by water based PET/CT scans

SECONDARY OUTCOMES:
24-hour blood pressure | Measured after each treatment period (day 6 and approximately day 26)
  Change in systolic 24-hour blood pressure
Vasoactive hormones | Measured after each treatment period (day 6 and approximately day 26)
  Change in plasma levels of angiotensin II, aldosterone, renin, brain natriuretic peptide (BNP), atrial natriuretic peptide (ANP), copeptin
Beta-hydroxybutyrate | Measured after each treatment period (day 6 and approximately day 26)
  Change ind p-beta-hydroxybutyrate
Renal tubular transport proteins | Measured after each treatment period (day 6 and approximately day 26)
  Urine excretions of aquaporin 2 (AQP2), thiazide-sensitive sodium-chloride cotransporter (NCC) and distal epithelial sodium channel (ENaC)

CONTACTS AND LOCATIONS:
Overall Officials: Jesper N Bech, PhD, Prof, Principal Investigator — University Clinic in Nephrology and Hypertension
Locations (1):
- The University Clinic of Nephrology and Hypertension, Herning, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No